CLINICAL TRIAL: NCT01644435
Title: A Prospective, Multicentric, Open Label, Bio Interventional, Phase I, Phase II Pilot Study to Evaluate the Safety and Efficacy of Autologous Human Platelet Lysate (HPL) for Treatment of Acne Scarring
Brief Title: A Pilot Study to Determine Safety & Efficacy of Autologous Human Platelet Lysate (HPL) in Treatment of Acne Scarring
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRPL/HPL-AS/11-12/004
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: ACNE SCARRING

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study arm A (Other): Subjects will receive a single injection of Autologous Human Platelet Lysate for acne scarring
  Interventions: Biological: Autologous Human Platelet Lysate
- Study arm B (Other): Subjects will receive two injections of Autologous Human Platelet Lysate at an interval of one month for acne scarring.
  Interventions: Biological: Autologous Human Platelet Lysate

INTERVENTIONS:
Biological: Autologous Human Platelet Lysate — Subjects will receive a single injection of Autologous Human Platelet Lysate for acne scarring
  Arms: Study arm A
Biological: Autologous Human Platelet Lysate — Subjects will receive two injections of Autologous Human Platelet Lysate at an interval of one month for acne scarring
  Arms: Study arm B

SUMMARY:
This is a multicentre, open label, randomized, pilot study to evaluate safety and efficacy of Human Platelet Lysate (HPL) in subjects with Acne Scarring. The study is being conducted at 2 centers in India. The primary endpoint is change in the Global Acne scarring classification scores from screening to end of the study. The secondary endpoints are Photographic Assessment, Physicians assessment score and Patients self assessment score.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male and female), aged 18 to 40 years (both inclusive).
* Subject willing to refrain from any other treatment of Acne Scarring during entire study duration.
* Non-pregnant, non-lactating females who agree to use adequate and acceptable methods of contraception from screening and throughout the course of the study.
* Subjects who are willing to give informed consent and adhere to the study protocol.

Exclusion Criteria:

* Subjects with active infection or active acne.
* Subjects receiving treatment: NSAIDs treatment within the last 7 days prior to the study.
* Subjects with history of connective tissue disease.
* Subjects with metabolic or hematopoietic disorders.
* Subjects with known bleeding disorders such as platelet dysfunction syndrome, thrombocytopenia, hypofibrinogenemia.
* Subjects who have received prior chemotherapy and radiotherapy
* Subjects unwilling to or unable to comply with the study protocol.
* Subjects taking concomitant therapy that might interfere with the study results in the investigator's opinion or participating in another trial in the past 30days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes in the Global Acne scarring classification | Day 0, End of study - Month 3

SECONDARY OUTCOMES:
Photographic Assessment | Day 0, Month 1, Month 2 End of study - Month 3

OTHER OUTCOMES:
Physician's assessment scores | End of Study - Month 3
Patient's assessment scores | End of Study - Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Patil, Dr., Principal Investigator — Dermocosmetic laser center hair and skin clinic; Pankaj Maniar, Dr., Principal Investigator — Radiance Cosmetology Clinique
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India